# Statistical Analysis Plan: TB006AD2102

Study Title: A Seamless Phase 1b/2a Double-blind, Randomized, Multiple

dose, Multi-center, Sequential Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics

and Efficacy of TB006 in Patients with Mild to Severe

Alzheimer's Disease

Study Number: TB006AD2102

**Study Phase:** Phase 1b/2a

**Sponsor:** TrueBinding, Inc.

300 Lincoln Center Drive

Suite 200

Foster City, CA

94404

**Version:** Final 2.0

NCT Number: NCT05074498

**Date:** 11Apr2022

# **Confidentiality Statement**

This document contains confidential and proprietary information, and is not to be distributed to any third party.



# 1. TABLE OF CONTENTS

| 1. T. | ABLE OF CONTENTS | 2 |
|---|---|---|
| LIST ( | OF TABLES | 2 |
| LIST ( | OF FIGURES | |
| LIST ( | OF APPENDICES | ∠ |
| 2. S | IGNATURE PAGE | 4 |
| 3. L | IST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
| 4. IN | NTRODUCTION | 10 |
| 5. T | RIAL OBJECTIVES | 10 |
| 5.1. | Primary Objectives | 10 |
| 5.2. | Secondary Objectives | 10 |
| 6. S | TUDY DESIGN CONSIDERATIONS | |
| 6.1. | Study Design | |
| 6.1.1. | Justification of Sample Size | |
| 6.2. | Efficacy Endpoints | |
| 6.3. | Safety Endpoints | 14 |
| 6.4. | Pharmacokinetic Endpoints | 15 |
| 6.5. | Pharmacodynamic Endpoints | 16 |
| 6.6. | Other Drug Related Endpoints | 16 |
| 7. S | TUDY POPULATIONS | 16 |
| 7.1. | Analysis Populations | 16 |
| 7.1.1. | Full Analysis Set (FAS) | 16 |
| 7.1.2. | Safety Analysis Set (SAS) | 16 |
| 7.1.3. | Pharmacokinetic Analysis Set (PKS) | 16 |
| 7.1.4. | Pharmacodynamic Analysis Set (PDS) | 16 |
| 7.1.5. | Efficacy Analysis Set – Part 2 (EAS2) | 17 |
| 7.2. | Subgroups | 17 |
| 8. C | HANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL | 17 |
| 9. O | VERALL STATISTICAL CONSIDERATIONS | 17 |
| 9.1. | General Conventions | 17 |
| 9.2. | Baseline definition | 18 |
| 9.3. | Handling of PK Concentration Values Below Lower Limit of Quantification | 18 |
| 9.4. | Handling of Missing Data | |
| 9.4.1. | Partial Dates | 19 |
| 9.4.2. | Missing Value Imputation for Efficacy Endpoints – Part 2 | 20 |
| 9.5. | MMRM Method | |
| 9.6. | Seriousness, Relationship and Severity of AEs | 20 |

| 9.7. | | |
|---|---|---|
| | Visit Windows/Unscheduled Visits | 21 |
| 10. S | TATISTICAL ANALYSIS METHODS | 21 |
| 10.1. | Subject Disposition | 21 |
| 10.2. | Demographics and Baseline Characteristics | 22 |
| 10.3. | Medical History And Viral Serology | 23 |
| 10.4. | Prior and Concomitant Medications and Procedures | 23 |
| 10.5. | Pharmacokinetics | 24 |
| 10.6. | Pharmacodynamics | 26 |
| 10.7. | Treatment Compliance and Exposure | 26 |
| 11. E | FFICACY PARAMETERS | 27 |
| 11.1. | Primary Analysis | 27 |
| 11.2. | Secondary Analysis | 27 |
| 11.2.1 | . Change from Baseline at Day 36 on the Clinical Dementia Rating Scale – Sum of Boxes Total Score | 27 |
| 11.2.2 | . Responder on the Clinical Dementia Rating Scale at Days 36 and 104 | 27 |
| 11.2.3 | . Change from baseline Cognitive Drug Research System Battery at Days 36 and 104 | 28 |
| 11.2.4 | . Change from baseline MMSE total score at Days 36 and 104 | |
| | . Change from baseline NPI total score at Days 36 and 104 | |
| 11.3. | Sensitivity Analysis | 28 |
| 11.4.1 | . Change From Baseline Through End of Study – Cognition Parameters | 28 |
| 11.5. | Interim Analysis | 29 |
| 11.5.<br>11.6. | Interim Analysis Subgroup Analyses | |
| 11.6. | j | 29 |
| 11.6. | Subgroup Analyses | 29 |
| 11.6.<br>12. S | Subgroup AnalysesAFETY AND TOLERABILITY | 29<br>30 |
| 11.6.<br>12. S<br>12.1. | Subgroup Analyses AFETY AND TOLERABILITY Adverse Events | 29<br>30<br>31 |
| 11.6.<br>12. S<br>12.1.<br>12.2. | Subgroup Analyses AFETY AND TOLERABILITY Adverse Events Laboratory Results | 29<br>30<br>31<br>33 |
| 11.6.<br>12. S<br>12.1.<br>12.2.<br>12.3. | Subgroup Analyses AFETY AND TOLERABILITY Adverse Events Laboratory Results Electrocardiogram (12-Lead) | 29<br>30<br>31<br>33 |
| 11.6.<br>12. S<br>12.1.<br>12.2.<br>12.3.<br>12.4.<br>12.5. | Subgroup Analyses AFETY AND TOLERABILITY Adverse Events Laboratory Results Electrocardiogram (12-Lead) Vital Signs | 29<br>30<br>31<br>33<br>35 |
| 11.6.<br>12. S<br>12.1.<br>12.2.<br>12.3.<br>12.4.<br>12.5. | Subgroup Analyses AFETY AND TOLERABILITY Adverse Events Laboratory Results Electrocardiogram (12-Lead) Vital Signs Columbia Suicide Severity Rating Scale | 29<br>30<br>31<br>35<br>35<br>36 |



| 13.3. Immur | ogenicity analysis |
|---|---|
| | NCES |
| | ICES38 |
| LIST OF T | ARIFS |
| LI31 OI 1 | ADLLO |
| Table 1. | Handling of Partial Dates |
| Table 2. | CTCAE Grades |
| Table 3. | ECG Measurements |
| Table 4. | Vital Sign Tests Performed35 |
| LICTOFF | ICURES |
| LIST OF F | IGURES |
| Figure 1 | Study Design and Treatment Schema for Part 1 and Part 2 |
| Figure 2. | Study Design and Treatment Schema – Interleave with Study TB006HV110113 |
| S | |
| LIST OF A | PPENDICES |
| Appendix I: | Schedule of Assessments and Procedures |
| Appendix II: | |
| | Summary of Laboratory Assays Performed |
| * * | Potentially Clinically Important Values |
| 1 1 P P 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 1 Overrount j Chimeent j himporeente vereente ve |




# 2. SIGNATURE PAGE

| Study Title: | A Seamless Phase 1b/2a Double-blind, Randomized, Multiple |
|---|---|
| v | dose, Multi-center, Sequential Dose-escalation Study to Assess |
| | the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics |
| | and Efficacy of TB006 in Patients with Mild to Severe |
| S - 1950 | Alzheimer's Disease |
| Study Number: | TB006AD2102 |
| Prepared by: Signing Time 053E504EE0 | con: I am the author of this document : 12-Apr-2022 03:33:33 EDT CB249B9B7E731AE1A775A71 PhD statistician, Biostatistics gs |
| Reviewed by: Senior Biostat MMS Holding | Date: Distriction II, Biostatistics Scon: I have reviewed this document on the common of the commo |
| Signing Time: | on: I approve this document 12-Apr-2022 10:07:35 PDT 6694A04A3393E173E8742DB PharmD lopment Lead |


# 3. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

ACR Assessment/Collection/Result

AD Alzheimer's Disease

ADA Anti-Drug Antibody

ADL Activities of Daily Living

AE Adverse Events

ALP Alkaline Phosphatase

ALT Alanine Aminotransferase

Anti-HBc IgM Hepatitis B Core Antibody

Anti-HCV Hepatitis C Antibody

ApoE4 Apolipoprotein E4

AR(1) Auto-regressive

AST Aspartate aminotransferase

ATC Anatomical Therapeutic Chemical

AUC $_{0-6}$  Area under the concentration time curve from time zero to the 6-hour

post end of infusion timepoint

AUC<sub>0-last</sub> Area Under the Concentration-Time Curve from Zero Time to the Last

Measurable Time Point

AUC<sub>tau</sub> Area Under the Concentration-Time Curve over a Dosing Interval

BLQ Below the Lower Limit of Quantification

BMI Body Mass Index

BUN Blood Urea Nitrogen

CDER Center for Drug Evaluation and Research

CDR Cognitive Drug Research

CDRS Clinical Dementia Rating Scale

CFB Change from Baseline

CI Confidence Interval

CL Total Clearance

cm Centimeter

C<sub>max</sub> Maximum Observed Plasma Concentration


TB006 Statistical Analysis Plan: TB006AD2102



CMH Cochran Mantel-Haenszel

COVID Coronavirus Disease

CPK Creatine Phosphokinase

CSF Cerebrospinal Fluid

C-SSRS Columbia Suicide Severity Rating Scale

CTCAE Common Terminology Criteria for Adverse Events

C<sub>trough</sub> Concentration at the End of a Dosing Interval

D Day

DBP Diastolic Blood Pressure

DSM 5 Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition

E/D Early Discontinuation

EAS2 Part 2 – Efficacy Analysis Set

ECG Electrocardiogram

eCRF Electronic Case Report Forms

FAS Full Analysis Set

FDA Food and Drug Administration

FSH Follicle-stimulating Hormone

HbA1c Hemoglobin A1c

HBsAg Hepatitis B Surface Antigen

hCG Human Chorionic-Gonatropin

HDL High-Density Lipoprotein

HIV Human Immunodeficiency Virus

IgM anti HBc Immunoglobulin M Antibody to Hepatitis B Core Antibody

IV Intravenously

Kg Kilogram

KR Kenward-Roger

LDL Low-Density Lipoprotein

LS Least Square


TB006

Statistical Analysis Plan: TB006AD2102



MAD Multiple Ascending Dose

MAR Missing at random

MCH Mean Corpuscular Hemoglobin

MCV Mean Corpuscular Volume

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed Model Repeated Measures

MMSE Mini-Mental State Examination

NCA Non-Compartmental Analysis

1 ton Compartmental I mary sis

NINCDS-ADRDA National Institute of Neurological and Communicative Disorders and

Stroke – Alzheimer's Disease and Related Disorders Association

NPI Neuropsychiatric Inventory

PCI Potentially Clinically Important

PCS Potentially Clinically Significant

PD Pharmacodynamics

PDS Pharmacodynamic Analysis Set

PK Pharmacokinetic

PKS Pharmacokinetic Analysis Set

PT Preferred Term

QTcB QT Corrected Interval Using Bazett equation

QTcF QT Corrected Interval Using Fridericia's Formula

qw Weekly

RBC Red Blood Cell

SAD Single Ascending Dose

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SAS Safety Analysis Set




SD Standard Deviation

SOC System Organ Class

SRC Safety Review Committee

t<sub>1/2</sub> Terminal Elimination Phase Half Life

TBL Total Bilirubin

TEAE Treatment-Emergent Adverse Event

t<sub>max</sub> Time at Which Maximum Plasma Concentration Occurs

TOEPH Heterogeneous Toeplitz

TSH Thyroid-Stimulating Hormone

ULN Upper Limit of Normal

UN Unstructured

V<sub>z</sub> Volume of Distribution

WHO DD World Health Organization-Drug Dictionary




# 4. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to describe the framework for the reporting, summarization and statistical analysis methodology of the safety, tolerability, pharmacokinetic (PK), pharmacodynamics (PD) and efficacy endpoints measured throughout the study. It is based on Protocol TB006AD2102 Amendment 2.0 dated 15 October 2021.

# 5. TRIAL OBJECTIVES

# **5.1. PRIMARY OBJECTIVES**

The study is planned to conduct in two different parts, and primary objectives for Part 1 are as listed:

- To determine the safety and tolerability of multiple doses of TB006
- To determine the PK profile of multiple doses of TB006
- To determine the maximum tolerated dose of multiple doses of TB006
- To assess the immunogenicity of TB006 (production of anti-TB006 antibody)

The primary objective for Part 2 is as follows:

• To determine the clinical efficacy of TB006 in patients with mild to severe Alzheimer's disease (AD)

# **5.2. SECONDARY OBJECTIVES**

There is no secondary objective planned for Part 1 of the study.

The following are the secondary objectives for the Part 2 of the study:

- To determine the clinical efficacy of TB006 in patients with mild to severe AD
- To determine the safety and tolerability of multiple doses of TB006
- To determine the PK following multiple doses of TB006




# 6. STUDY DESIGN CONSIDERATIONS

# **6.1. STUDY DESIGN**

This is a seamless, two-part Phase 1b/Phase 2a, multi-center, randomized, double-blind, placebo-controlled study. Part 1 is a multiple ascending dose (MAD) escalation study to evaluate the safety, tolerability, PK, PD, and efficacy of TB006 in patients with AD. Part 2 is a multi-center, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy of TB006 after 1 month of treatment. The total study duration for each patient will be up to approximately 19 weeks.

Patients will receive a total of 5 doses, given in qw intervals. In Part 1, the planned starting dose in Group 1 will be 140 mg qw for 5 weeks. Subsequent planned doses are 420 and 1,000 mg qw for Groups 2 and 3, respectively. The planned dose in Part 2 will be the highest safe and well-tolerated dose from Part 1. All doses are infused IV over 1 hour. Part 1 will interleave with the single ascending dose (SAD) study (Study TB006HV1101). Each group in Part 1 will commence after the safety, tolerability, and PK of the single dose equivalent to the combined total of 5 qw doses planned in this study has been established. Explicitly, dosing in Group 1 (140 mg qw) will commence when the safety and tolerability of the 700 mg single dose in the SAD study has been established. Groups 2 (420 mg qw) and 3 (1000 mg qw) will begin after a review of the available safety, tolerability, and PK data from the previous group; and after the 2,100 and 5,000 mg single dose, respectively, has been administered. Dose levels may be adjusted depending on the safety, tolerability, and available PK of doses in the SAD study and previous groups in this study. Patients will be enrolled across all active centers into each dose group sequentially.

In Part 1, 8 patients will be enrolled into each dose group; 6 patients in each group will be randomized to active TB006 treatment, and 2 patients to placebo.

Dose escalation decisions will use safety, tolerability, and available PK data through the first dose administered to the last patient in each group and a minimum of 14 days from the respective dose group that has been dosed in the SAD study (Protocol number TB006HV1101). Data will be reviewed by a blinded Safety Review Committee (SRC).

Part 2 will commence after the last patient in Part 1 has received their first dose. The planned dose in Part 2 will be 1,000 mg qw  $\times$  5 doses, but may be adjusted depending on the safety and tolerability of the doses in Part 1. Patients will be randomized to active TB006 or placebo (1:1) and will follow the same dosing schedule and procedures (with some exceptions – see Part 2 schedule of assessment) as in Part 1. Randomization in Part 2 will be stratified according to baseline patient severity, with mild AD patients [Mini-Mental State Examination (MMSE) 21-24] and moderate-severe AD patients (MMSE  $\leq$  20) in each stratum.

This is an outpatient study. Patients will return to the clinic for screening and baseline procedures, on dosing days, and on follow-up visits. Patients will have the option of checking into the clinic and staying overnight on Day -2 or Day -1, as well as on days prior to the other dosing days.

Assessments for safety and tolerability, efficacy, PK, and PD are performed throughout the study. If a patient reports any adverse events (AEs), they may be required to return to the clinical




unit at the discretion of the investigator for additional assessments. All AEs must be followed to adequate resolution.

Figure 1 Study Design and Treatment Schema for Part 1 and Part 2



<sup>\*</sup> Study drug administration

Note: Visit days and procedures will occur during a window of  $\pm$  2 days from Day 1 to End of Treatment. D = Day; IV = intravenously, qw = weekly.






Dosing in Group 1 (140 mg TB006/placebo aww) will commence when the safety and tolerability of the 700 mg single dose in the SAD study has been established. Groups 2 (420 mg TB006/placebo qw) and 3 (1,000 mg TB006/placebo qw) will begin after a review of the available safety, tolerability and PK data from the previous group; and after the 2,100 and 5,000 mg, respectively, have been administered.

\* Study drug administration

Note: Visit days and procedures will occur during a window of  $\pm\,2$  days from Day 1 to End of Treatment

D = Day; IV = intravenously; PK = pharmacokinetic; qw = weekly; SAD = single ascending dose.




# **6.1.1.** JUSTIFICATION OF SAMPLE SIZE

In Part 1, patients will be recruited sequentially in separate increasing dose groups, with each group randomizing 6 patients to a specific dose of TB006 and 2 randomized to placebo. If all 3 planned dose levels are investigated, the study will recruit approximately 24 patients in total (18 receiving TB006 treatment at the different dose levels, and 6 receiving placebo).

In Part 2, patients will be randomized to TB006 or placebo in a 1:1 ratio so that approximately 58 patients will be randomized to each group. Randomization in Part 2 will be stratified according to baseline patient severity, with mild AD patients (MMSE 21-24) and moderate-severe AD patients (MMSE  $\leq$  20) in each stratum. Patients enrolled at the same TB006 dose level in Part 1, as well as all placebo patients, will be included in the efficacy analyses in Part 2. Thus, the number of patients in each group for the primary efficacy analysis will be approximately 64.

Assuming that the standard deviation (SD) of change from baseline (CFB) Clinical Dementia Rating Scale (CDRS) - Sum of Boxes at Day 104 is 0.5, a total of 128 patients will provide 80% power to detect a mean CFB difference of 0.25 at Day 104 using a 2-sided, 2 sample t-test at the 5% level of significance.

# **6.2. EFFICACY ENDPOINTS**

For Part 1, there is no efficacy endpoint planned for primary and secondary analysis, but following endpoints is planned for exploratory analysis:

- CFB through end of study on the CDRS Sum of Boxes total score
- CFB through end of study on the Cognitive Drug Research (CDR) System Battery Score, composite scores, and individual task measures
- CFB through end of study on the MMSE score
- CFB through end of study on the Neuropsychiatric Inventory (NPI) score

For Part 2, the planned primary efficacy endpoint is:

• CFB through Day 104 on the CDRS – Sum of Boxes total score.

And the associated secondary endpoints are as under:

- CFB through Day 36 on the CDRS Sum of Boxes total score
- Proportion of responders on the CDRS Sum of Boxes at Days 36 and 104
- CFB to Days 36 and 104 on the CDR System Battery, composite scores, and individual task measures
- CFB to Days 36 and 104 on the MMSE score
- CFB to Days 36 and 104 on the NPI score

# **6.3. SAFETY ENDPOINTS**

The safety endpoints for Part 1 and Part 2 of the study will be recorded and reported throughout the safety reporting period. The safety reporting period is from Day 1 (start of TB006 infusion) through Day 104. Safety endpoints for both protocol parts of this study include:

• Incidence of AEs and serious adverse events (SAEs)




- Clinical Safety Laboratory Assessments
- Vital Signs
- Electrocardiograms
- Suicidal Ideation and Behavior Risk Monitoring
- Physical and Neurological Examinations

The safety endpoints listed above will be reported as primary endpoints for Part 1 of the study and as secondary endpoints for Part 2 of the study.

# **6.4. PHARMACOKINETIC ENDPOINTS**

The PK analysis will be performed using PK parameters derived by non-compartmental analysis (NCA) using the TB006 plasma concentration time data. The PK parameters will be estimated using actual sampling time relative to the start of infusion.

For Part 1 of the study, the PK analysis will be performed as primary endpoint and includes, but not limited to:

- Area under the concentration time curve from time zero to the 6-hour post end of infusion timepoint (AUC<sub>0-6</sub>) (Days 1, 8, and 29)
- Area under the concentration time curve over a dosing interval (AUC<sub>tau</sub>) (Days 1 and 29)
- Area under the concentration-time curve from zero time to the last measurable time point (AUC<sub>0-last</sub>) (Day 29)
- Maximum observed plasma concentration (C<sub>max</sub>) (Days 1, 8, and 29)
- Time at which maximum plasma concentration occurs  $(t_{max})$  (Days 1, 8, and 29)
- Concentration at the end of a dosing interval (C<sub>trough</sub>) (Days 8, 15, 22, 29, and 36)
- Terminal elimination phase half-life (t½) (Day 29 only)
- Total clearance (CL), calculated as dose/AUC<sub>tau</sub>. (Day 29 only)
- Volume of distribution (V<sub>z</sub>), calculated as dose/kel × AUC<sub>tau</sub>, where kel is the apparent elimination rate-constant, computed by log linear regression of the terminal log linear segment of the plasma concentration versus time curve (Day 29 only).

The extent of CSF distribution as estimated by TB006 CSF concentrations on Day 36 will also be determined.

For Part 2 of the study, the PK analysis will be performed as secondary endpoint and will include:

- Maximum observed plasma concentration (C<sub>max</sub>) (Days 1, 8, and 29)
- Concentration at the end of a dosing interval (C<sub>trough</sub>) (Days 29 and 36)
- Area under the concentration-time curve from zero time to the last measurable time point (AUC<sub>0-last</sub>) (Day 29)
- Terminal elimination phase half-life (t<sub>1/2</sub>) (Day 29 only)

Note that no CSF will be collected in Part 2 of the study.




6.5. PHARMACODYNAMIC ENDPOINTS

# **6.6. OTHER DRUG RELATED ENDPOINTS**

Apart from above analysis, following other drug related assessment will also be performed for Part 1, secondary analysis, of the study.

- Assessment of maximum tolerable dose
- Detection of anti-TB006 antibodies (from PK plasma sampling)

# 7. STUDY POPULATIONS

# 7.1. ANALYSIS POPULATIONS

# 7.1.1. FULL ANALYSIS SET (FAS)

The Full Analysis Set (FAS) includes all subjects who are randomized to study drug. The FAS will be used for the analysis of disposition and protocol deviations.

# 7.1.2. SAFETY ANALYSIS SET (SAS)

The Safety Analysis Set (SAS) includes all subjects in the FAS who received at least one dose of study drug. Subjects in this analysis set will be analyzed according to the study drug they actually received. The FAS and the SAS will be the same if all randomized patients are dosed with study drug. The SAS will be used for all analyses, except for disposition, protocol deviations, PK and PD.

# 7.1.3. PHARMACOKINETIC ANALYSIS SET (PKS)

The Pharmacokinetic Analysis Set (PKS) includes all subjects who received assigned dose of TB006 and have at least one post-dose blood sample with measurable TB006 concentrations. The PKS will be used for all PK analyses.

# 7.1.4. PHARMACODYNAMIC ANALYSIS SET (PDS)

The Pharmacodynamic Analysis Set (PDS) includes all subjects who received assigned dose of TB006 or placebo and have at least one post-dose evaluable PD assessment. The PDS will be used for all PD and efficacy analyses.


# 7.1.5. EFFICACY ANALYSIS SET – PART 2 (EAS2)

The Part 2 – Efficacy Analysis Set (EAS2) includes all subjects who received assigned dose of TB006 in Part 2 and the subjects enrolled at the same TB006 dose level in Part 1, as well as all placebo patients will be included and have at least one post-dose evaluable PD assessment across subject. The EAS2 will be used for all efficacy analysis planned for Part 2 of the study.

#### 7.2. SUBGROUPS

The dispositions, efficacy, PK/PD, biomarker, and immunogenicity analysis for Part 2 will be presented for overall and baseline patient severity: mild AD patients (MMSE 21-24) and moderate-severe AD patients (MMSE  $\leq$  20).

# 8. CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL

The following analyses described in this SAP are not mentioned in the study protocol:

• Assessment of dose proportionality (see Section 10.5: Pharmacokinetics).

# 9. OVERALL STATISTICAL CONSIDERATIONS

# **9.1. GENERAL CONVENTIONS**

Summary statistics will be presented for categorical data as number and percentage [n (%)] where the percentage is displayed to one decimal point (e.g., 98.1).

Descriptive statistics will be presented for continuous data with applicable decimal precision as follows in relation to the source data (indicated as N), with a maximum of three decimals to be displayed:

- Number (n).
- Mean, (N+1).
- SD, (N+2).
- Median, (N+1).
- Minimum, (N+0).
- Maximum, (N+0).




Study day is calculated relative to the first dose of study drug infusion and will thus in most cases coincide with the visit naming (e.g., Day 1 will be on study day = 1, Day 15 will be on study day = 15 etc.)

• If the current assessment/collection/result (ACR) date is on or after first dose of study drug infusion:

$$Study Day = (Current ACR Date - First dose of Study Drug infusion Date) + 1$$

• If the current ACR date is before first dose of study drug infusion:

$$Study Day = (Current ACR Date - First dose of Study Drug Infusion Date)$$

Study day will not be calculated if either the current ACR or the first dose of study drug infusion date is incomplete or missing.

All the tables in Part 1, will be displayed by treatment groups (i.e., TB006 140 mg qw, TB006 420 mg qw, TB006 1000 mg qw, and Pooled placebo).

The dispositions, efficacy, PK/PD, biomarker, and immunogenicity analysis for Part 2 will be classified by treatment groups (i.e., TB006 and Placebo) and baseline AD severity stratifications [i.e. mild AD (MMSE 21-24) and moderate-severe AD (MMSE  $\leq$  20)]. For efficacy tables of Part 2, the subjects enrolled at the same TB006 dose level in Part 1, as well as all placebo patients will be included.

For all baseline, safety and efficacy assessments, the subjects will be tabulated using the actually received treatment. For example, if there is a subject who is planned to receive TB006 but accidentally gets treated with one of the other regimens, the subject will be tabulated under the other regimen actually received.

The tables and listing for both protocol parts will be presented separately. The detailed layout will be presented in mock shell.

# 9.2. BASELINE DEFINITION

Baseline is defined as the last available value prior to the subject receiving first dose of study drug infusion (i.e., Day 1). If the potential Baseline ACR is on Day 1 (and time is not recorded), it is assumed that the ACR occurred before the start of first dose of study drug infusion.

CFB is calculated as:

$$CFB = Observed value - Baseline Value$$

Percentage change from Baseline (CFB%) is calculated as:

$$CFB\% = (CFB \div Baseline\ Value) \times 100$$

# 9.3. HANDLING OF PK CONCENTRATION VALUES BELOW LOWER LIMIT OF QUANTIFICATION

For PK concentrations, values that are below the lower limit of quantification (BLQ) the following handling measures will be applied:




- For NCA, pre-dose concentrations prior to the first dose of TB006 that are BLQ will be set to zero. Post-dose concentrations that are BLQ and occur before the first quantifiable concentration will also be treated as zero. Post-dose concentrations that are BLQ but occur after the first quantifiable concentration will be treated as missing.
- For summary statistics, BLQ concentrations will be treated as zero.
- In listing presentation these values will be marked/footnoted as being BLQ.

#### 9.4. HANDLING OF MISSING DATA

No formal imputation of missing data is planned for Part 1 of the study. There are however a few handling conventions and assumptions applicable to partial/missing data points which are described in the following subsections.

# 9.4.1. PARTIAL DATES

Although partial dates will not be 'filled up' in this study, some assumptions will be made in regards partial dates for background calculation/classification purposes as appropriate (for AEs, prior/concomitant medications etc.)

Table 1. Handling of Partial Dates

| Parameter | Missing | Additional Conditions | Imputation |
|---|---|---|---|
| Start date | D | M and Y same as M and Y of first dose of study drug | Date of first dose of study drug |
| | | M and/or Y not same as date of first dose of study drug | First day of month |
| | D and M | Y same as Y of first dose of study drug | Date of first dose of study drug |
| | | Y prior to Y of first dose of study drug<br>but same as Y of screening date | Date of screening date |
| | D, M and Y | None - date completely missing | Date of first dose of study drug |
| Stop date | D | M and Y same as M and Y of last dose of study drug | Date of last dose of study drug |
| | | M and/or Y not same as date of last<br>dose of study drug | Use last day of month |
| | D and M | Y same as Y of last dose of study drug | Date of last dose of study drug |
| | | Y not same as Y of last dose of study drug | Dec 31 |
| | D, M and Y | None - date completely missing | No imputation, but assume ongoing |

D = day, M = month, Y = year

Note: In all cases, if an estimated start date is after a complete stop date, use the first day of the stop date month.

Similarly, if the estimated stop date is before a complete or imputed start date, use the last day of the start day month.

In all cases, if it cannot be determined if the AE/medication occurred prior to or after the first dose of study drug infusion, the AE should be defined as treatment emergent, and medication will be considered as concomitant medication.




# 9.4.2. MISSING VALUE IMPUTATION FOR EFFICACY ENDPOINTS - PART 2

Apart from handling conventions and assumptions applicable to partial/missing data points mentioned above, there will be additional imputation for missing efficacy assessments listed under:

- CDRS Sum of Boxes total score
- MMSE score
- NPI score

For these imputations, the missingness will be considered as missing at random (MAR). There will be no imputation for individual missing values, but missing data will be imputed implicitly using Mixed Model Repeated Measures (MMRM).

The MMRM analysis will be performed for above listed efficacy endpoints as described in Section 9.5.

# 9.5. MMRM METHOD

The primary and secondary efficacy endpoints associated with efficacy assessments listed in Section 9.4.2 will be analyzed using a MMRM model. The model will include treatment group, visit, stratification factor (MMSE  $\leq$  20 and 21-24), and treatment by visit as fixed effects and associated baseline assessment as covariate. The model will use visit as repeated component in the model.

An unstructured (UN) covariance structure will be applied for the MMRM. In the event the UN covariance matrix results in non-convergence of the model, then the Heterogeneous Toeplitz (TOEPH) and auto regressive [i.e. AR(1)] covariance structures will be used, respectively, with separate subject random effect. The Kenward-Roger (KR) approximation will be used to estimate denominator degrees of freedom.

The least square (LS) mean for CFB and associated 95% confidence interval (CI), and standard error will be presented for each treatment group.

The MMRM model will utilize all available data values for respective efficacy assessments.

# 9.6. SERIOUSNESS, RELATIONSHIP AND SEVERITY OF AES

Missing seriousness, severity and relationship of AEs that have been queried and remain missing after such, will be treated 'worst case' for presentation filtering purposes as follows:

- Missing seriousness: Will be considered as serious and included in the SAE displays.
- Missing relationship: Will be considered as related and included in the related AE displays.
- Missing severity:
  - o If subject has died, will be considered as Grade 5 severity across all associated displays.




- o If subject has not died but subject had intervention indicated for the AE, will be considered as Grade 4 severity across all associated displays.
- o If none of the previous conditions are met, will be considered as Grade 3 severity across all associated displays.

# 9.7. VISIT WINDOWS/UNSCHEDULED VISITS

No mapping/renaming of visits (unscheduled or otherwise) will be done for this study. That is, only regular scheduled visit data will be used for summarization in tables. However, all collected data will be listed.

Unscheduled visits will be considered eligible for Baseline values. Unscheduled visit results will also be considered eligible for testing of potentially clinically significant (PCS) values (laboratory, Electrocardiogram (ECG) and vital signs).

# **10.STATISTICAL ANALYSIS METHODS**

#### **10.1.** SUBJECT DISPOSITION

The following disposition related items are planned to be listed using the protocol part and analysis set indicated in parentheses:

- Screening failures (Part 1 All subjects)
- Screening failures (Part 2 All subjects)
- Randomized subjects (Part 1 FAS)
- Randomized subjects (Part 2 FAS)
- Unblinded subjects, if any (Part 1 FAS)
- Unblinded subjects, if any (Part 2 FAS)
- Inclusion/Exclusion violations (Part 1 FAS)
- Inclusion/Exclusion violations (Part 2 FAS)
- Subject completion/discontinuation information (Part 1 FAS)
- Subject completion/discontinuation information (Part 2 FAS)
- Subject analysis set inclusions (Part 1 FAS)
- Subject analysis set inclusions (Part 2 FAS)
- Subject deviations (Part 1 FAS)
- Subject deviations (Part 2 FAS)

The following disposition related items are planned to be tabulated using summary and descriptive statistics as applicable, by treatment groups and baseline AD severity stratifications (for Part 2 only), using the protocol part and analysis set indicated in parentheses:




- Subject completion/discontinuation information (Part 1 All subjects). Including breakdown by reason for subject discontinuation.
- Subject completion/discontinuation information (Part 2 All subjects). Including breakdown by reason for subject discontinuation.
- Subject analysis set inclusions (Part 1 All subjects). Including reason for exclusion from analysis set, if required.
- Subject analysis set inclusions (Part 2 All subjects). Including reason for exclusion from analysis set, if required.
- Subject deviations (Part 1 FAS).
- Subject deviations (Part 2 FAS).

The data for these presentations are obtained from the following electronic Case Report Forms (eCRFs):

- Informed Consent
- Screen Failure
- Inclusion Exclusion Criteria
- Randomization
- End of Study

# 10.2. DEMOGRAPHICS AND BASELINE CHARACTERISTICS

The following demographics and baseline characteristic items will be listed using SAS for both protocol parts:

- Subject demographics:
  - o Age
  - o Sex
  - o Race
  - o Ethnicity
- Baseline vital characteristics:
  - o Height (cm)
  - Weight (kg)
  - $\circ$  BMI (kg/m<sup>2</sup>)
- Substance usage, including checking for:
  - o Tobacco/nicotine use
  - Alcohol use
  - o Drug use


The above demographic, baseline characteristics and substance use items are planned to be tabulated using summary and descriptive statistics as applicable, by treatment groups for SAS.

The data for these presentations will be obtained from the following eCRFs:

- Demography
- Physical Examination (for baseline height/weight)
- Medical History (for substance usage medical history)
- Drug and Alcohol Screening

The following items will be derived:

• Body mass index (BMI) at Baseline:

Baseline BMI = Baseline weight (kg)  $\div$  [Baseline height (m)]<sup>2</sup>

# 10.3. MEDICAL HISTORY AND VIRAL SEROLOGY

The medical history terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.1, Sep 2019.

The following medical history and viral serology baseline characteristic items will be listed using SAS for both protocol parts:

- Medical history:
  - Medical conditions or allergies reported
- Viral serology
  - o HBsAg
  - o IgM anti HBc
  - o anti HCV
  - o HIV
- COVID-19 status

The above medical history is planned to be tabulated using summary statistics, by treatment groups using SAS.

The data for these presentations will be obtained from the following eCRFs and external data:

- Medical History
- Viral Serology
- Laboratory Data

# 10.4. PRIOR AND CONCOMITANT MEDICATIONS AND PROCEDURES

A prior medication or procedure is defined as having started and ended prior to first dose of study drug infusion. Conversely, a concomitant medication or procedure is defined as either having started prior to first dose of study drug infusion and ended on/after first dose of study




drug infusion, is ongoing at Baseline or, having started on/after first dose of study drug infusion. Medications will be coded using the World Health Organization-Drug Dictionary (WHO-DD) Global Sep 2019 B3/C3 format.

Listings of prior and concomitant medications/procedures will be presented for both protocol parts as recorded in the eCRF (SAS).

Summary tables by WHO-DD Anatomical Therapeutic Chemical (ATC) level 3 and preferred name will be presented, by treatment groups on the following items:

- Prior medications/procedures (Part 1 SAS).
- Prior medications/procedures (Part 2 SAS).
- Concomitant medications/procedures (Part 1 SAS)
- Concomitant medications/procedures (Part 2 SAS)

The data for these presentations will be obtained from the Concomitant Medications Details eCRF.

The Prior/Concomitant status will be derived using the medication start and stop dates as per definition provided at the start of this section. For partial dates see Section 9.4.1.

#### **10.5. PHARMACOKINETICS**

The following PK listings are planned for presentation (PKS) for both protocol parts:

- TB006 plasma concentration levels
- TB006 CSF concentration level (Part 1 only)
- Pharmacokinetic parameters of plasma TB006
- Dose-normalized plasma exposure PK parameters (AUCs and  $C_{max}$ ) (Part 1 only).

The following descriptive summary tables are planned to be presented for subjects who received TB006 (PKS), by treatment groups and baseline AD severity stratifications (for Part 2 only):

- Plasma concentration of TB006 at each time points
- CSF concentration of TB006 at each time points (Part 1 only)
- Plasma PK parameters
- Dose-normalized exposure PK parameters (AUCs and C<sub>max</sub>) (Part 1 only, Days 1, 8, and 29, as applicable)
- Power model slope estimate for dose proportionality assessment (including 95% CI) (Part 1 only)

Figures of the following PK items are planned for presentation (PKS) for both protocol parts:

 Overlaid individual plasma concentration versus time plots (linear and semi-logarithmic scale) by treatment groups




- Overlaid mean plasma concentration versus time plots, presented by treatment groups (linear scale with and without SD)
- Overlaid mean plasma concentration versus time plots, presented by treatment groups (semi-logarithmic scale with and without SD)
- Boxplots of dose-normalized PK parameters (AUCs and C<sub>max</sub>), grouped by treatment groups grouped within each figure (Part 1 only, Days 1, 8, and 29, as applicable)
- Scatterplots of PK parameters (AUCs and C<sub>max</sub>), versus dose (as part of power model results), by treatment groups (Part 1 only, Days 1, 8 and 29, as applicable)

Assessment of dose proportionality will be performed by PK Day (Day 1, 8, and 29, as applicable) and will not be based strictly on statistical rule criteria but rather, several factors will be taken into account when assessing dose proportionality, such as:

- Power model results (e.g., the slope estimate and the width of the 95% CIs)
- Graphical evaluation (box plots of dose normalized AUCs and C<sub>max</sub>)
- Descriptive statistics by treatment groups of dose-normalized PK parameters

Evaluations of the dose proportionality of these parameters will include using the Power Model if there will be at least 3 dose levels available. A statistical linear relationship between the Intransformed PK parameters and the In-transformed dose will be fitted by using a mixed model with In-transformed dose as a covariate and random effect for intercept and subject. Here, (In-) stands for natural logarithm. Additional predictors may be included in the model. The general form of the Power Model is described as:

$$Ln(Y) = \beta_0 + \beta Ln(Dose) + \varepsilon$$

Where, Y represents the PK parameter (AUCs and  $C_{max}$ ), and  $\beta_{\theta}$  is constant. This approach is usually referred to as a power model because after exponentiation:

$$Y = \alpha \, (Dose)^{\beta}$$

Note that  $\beta = 1$  would correspond to perfect dose proportionality.

The following example SAS® code can be utilized and modified as needed:

```
Proc Mixed Data = <Dataset>;
   Class <subjectnum>
   Model <InY> = <InDose> / ddfm=kr;
   Random <intercept> / subject = <subjectnum> type=UN;
   Estimate 'Logdose - 1 unit' <Indose> 1/cl alpha=0.05;
   ods output estimates = <estimate>;
Run;
```

Where *<Dataset>* is the input dataset, *<subjectnum>* is the subject number, *<LnY>* is Ln(Y) (Y being the PK parameter in question, *<LnDose>* is Ln(Dose), *<intercept>* is the intercept and *<estimate>* is the output dataset containing the estimate.

The data for these presentations will be obtained from the external PK laboratory data and eCRF.






Descriptive summary tables of biomarker levels from both plasma and CSF (for Part 1 only) collection will be presented, by treatment groups and baseline AD severity stratifications (for Part 2 only), using PDS for both protocol parts, including CFB and CFB% through end of study.

The relationship between dose, Day 29 plasma TB006 PK exposure parameters (AUC<sub>tau</sub> and C<sub>max</sub>), Day 36 CSF TB006 concentration and PD biomarkers listed in Section 10.6 will be assessed graphically. Scatter plots of CFB and CFB% will be presented next to another in grid format for PD endpoint values versus TB006 AUC<sub>tau</sub> and  $C_{max}$ . The PD endpoints will be for timepoints Day 36 and end of study. The main measure of interest for consideration will be the CFB of PD biomarkers.

The data for these presentations will be obtained from the external laboratory data and eCRF.

# **10.7.**TREATMENT COMPLIANCE AND EXPOSURE

A listing of subject exposure to all the doses of TB006 will be presented including the date/time of dose and dose level exposed to (SAS) for both protocol parts separately. Also, the treatment compliance information will be listed.

A table containing summary statistics of dose level exposure, by treatment groups will also be presented using SAS.

Treatment compliance is defined as the number of IV doses (including partial doses, active and placebo) actually received divided by the number of doses expected (× 100) over the time period defined by the first infusion date and the last dose date.

Descriptive statistics for treatment compliance and the number and percentage of subjects with at least 80% compliant will be presented using SAS.

The data for these presentations will be obtained from the Study drug infusion eCRF.




# 11. EFFICACY PARAMETERS

All the efficacy analysis planned for Part 1 will be performed using PDS and efficacy analysis planned for Part 2 will be performed using EAS2. The EAS2 include all PDS subjects of Part 2, placebo subjects of Part 1 and subjects with same dose level in Part 1 pooled together.

# 11.1.PRIMARY ANALYSIS

There is no primary efficacy analysis planned for Part 1.

For Part 2, the CFB through Day 104 on the CDRS – Sum of Boxes total score is primary efficacy endpoint, and it will be analyzed using MMRM with treatment group, randomization strata (MMSE  $\leq$  20 and 21-24), visit, and treatment group (treated vs. placebo) by visit interaction as fixed effects and a baseline CDRS - Sum of Boxes score as a covariate. The LS mean difference, the 95% CI of the difference, and the p-value will be presented as well as the descriptive statistics.

#### 11.2. SECONDARY ANALYSIS

There is no secondary efficacy analysis planned for Part 1.

For Part 2, the following secondary analysis are planned.

# 11.2.1. CHANGE FROM BASELINE AT DAY 36 ON THE CLINICAL DEMENTIA RATING SCALE — SUM OF BOXES TOTAL SCORE

The secondary efficacy endpoint, CFB at Day 36 on the CDRS – Sum of Boxes, and will be analyzed and reported as described for the primary analysis in Section 11.1.

Also, the summary statistics will be tabulated for CDRS individual scores, sum of box total score and Global CDRS score by treatment groups and baseline AD severity stratifications.

#### 11.2.2. RESPONDER ON THE CLINICAL DEMENTIA RATING SCALE AT DAYS 36 AND 104

A responder is defined as at least 1-point improvement from baseline on the Sum of Boxes score. The patients with missing data will be included in the denominator and treated as a non-responder.

The proportion of the responders between treatment groups will be tested using the Cochran Mantel-Haenszel (CMH) test, adjusting for randomization strata (MMSE  $\leq$  20 and 21-24) and the common risk difference and the 95% CI will be presented.

Also, the number and percentages of responders over time will be tabulated by treatment groups and baseline AD severity stratifications.

The CDRS individual scores, sum of box total score, Global CDRS score and responder status will be listed as well.




# 11.2.3. CHANGE FROM BASELINE COGNITIVE DRUG RESEARCH SYSTEM BATTERY AT DAYS 36 AND 104

This endpoint is analyzed separately, and detail of analysis is described in CDR system battery SAP [5].

#### 11.2.4. CHANGE FROM BASELINE MMSE TOTAL SCORE AT DAYS 36 AND 104

The secondary efficacy endpoint, CFB at Day 36 and Day 104 on the MMSE total score will be analyzed using MMRM with treatment group, visit, and treatment group by visit interaction as fixed effects and a corresponding MMSE total baseline score as a covariate. The LS mean difference, the 95% CI of the difference, and the p-value will be presented as well as the descriptive statistics.

Also, the summary statistics will be tabulated for MMSE score by treatment groups and baseline AD severity stratifications.

The MMSE scores will be listed as well.

# 11.2.5. Change from Baseline NPI Total score at Days 36 and 104

The secondary efficacy endpoint, CFB at Day 36 and Day 104 on the NPI total score will be analyzed using MMRM with treatment group, randomization strata (MMSE  $\leq$  20 and 21-24), visit, and treatment group by visit interaction as fixed effects and a corresponding NPI total baseline score as a covariate. The LS mean difference, the 95% CI of the difference, and the p-value will be presented as well as the descriptive statistics.

Also, the summary statistics will be tabulated for NPI by treatment groups and baseline AD severity stratifications.

The individual and composite NPI scores will be listed as well.

#### 11.3. SENSITIVITY ANALYSIS

Not applicable for either part of this study.

# 11.4.1. CHANGE FROM BASELINE THROUGH END OF STUDY — COGNITION PARAMETERS

The observed and change/shift from baseline in results from the cognition parameters - CDRS individual scores, sum of box total score, Global CDRS score, Responders for CDRS-sum of boxes total score, MMSE score, and NPI total score will be summarized by treatment groups using continuous and categorical descriptive statistics.

The assessment associated with cognition parameters - CDR system battery, will be analyzed separately, and detail of analysis is described in CDR system battery SAP [5].






# 11.5.INTERIM ANALYSIS

No formal interim analysis planned for this study.

A SRC will meet for each dose cohort before continuing to the next dose cohort.

# 11.6.SUBGROUP ANALYSES

The subgroup analysis for Part 2 will be performed as described in Section 7.2.




# 12.SAFETY AND TOLERABILITY

#### **12.1.ADVERSE EVENTS**

The following AE definitions are applicable to both protocol parts of this study:

- AE reporting period: Defined from start of first dose of study drug infusion on Day 1 up to and including End of Study.
- AE: Any untoward medical occurrence in a subject.
- Treatment-emergent AE (TEAE): Defined as any AE that started on or after first dose of study drug infusion within the studies' AE reporting period.
- SAE: Defined as any AE that is indicated as serious on the AEs Details eCRF, as per investigator's assessment.
- Related AE: Defined as any AE that is indicated as related to study drug on the AEs Details eCRF, as per investigator's assessment.
- AE leading to discontinuation: Defined as any AE that has an "other action taken" indicated as "withdrawn from study" on the AEs Details eCRF.

All AEs will be coded using the MedDRA version 22.1, Sep 2019. The following AE items will be listed separately for each protocol parts using the SAS:

- All AEs
- AEs leading to study discontinuation
- Serious AEs
- AEs leading to death (if applicable)

The following items are planned to be presented in summary tables showing event incidence and corresponding subject count, experiencing said AE/AE type using the SAS, by treatment groups using SAS:

- AE overview, including row items for frequency of subjects [n(%)] experiencing:
  - o At least one AE
  - o AEs by toxicity grade
    - Grade 1
    - Grade 2
    - Grade 3
    - Grade 4
    - Grade 5
  - Serious AEs




- Related AEs
- Non-related AEs
- AEs leading to study discontinuation
- AEs leading to death
- AEs by system organ class (SOC) and preferred term (PT)
- AEs by descending incidence of PT
- AEs by toxicity grade (Common Terminology Criteria for Adverse Events [CTCAE] grading)
- Related AEs by SOC and PT
- Related AEs by descending incidence of PT.
- Serious AEs
- AEs resulting in death
- AEs leading to study discontinuation

Only TEAEs will be used for summarization of all tables, but for listing all AEs will be counted. The TEAE status will be derived using the AE start and stop dates as per definition provided at the start of this section. For partial dates see Section 9.4.1.

The data for these presentations will be obtained from the Adverse Events Details eCRF.

AE assignment to CTCAE toxicity grades is explained in Table 2 below.

Table 2. CTCAE Grades

| Grade | Grade Description | Grade Details |
|---|---|---|
| Grade 1 | Mild | Asymptomatic or mild symptoms; clinical or diagnostic observations only intervention not indicated |
| Grade 2 | Moderate | Minimal, local, or non-invasive intervention indicated, limiting age-<br>appropriate instrumental ADL* |
| Grade 3 | Severe | Severe or medically significant but not immediately life-threatening;<br>hospitalization or prolongation of hospitalization indicated; disabling;<br>limiting selfcare ADL* |
| Grade 4 | Life-threatening | Life-threatening consequences: urgent intervention indicated |
| Grade 5 | Fatal | Death related to AE |

ADL: activities of daily living.

# 12.2.LABORATORY RESULTS

In the context of this study the difference between potentially clinically important (PCI) and PCS results are defined as follows:


<sup>\*</sup>Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

<sup>\*\*</sup> Self-care ADL refer to bathing, dressing, and undressing, feeding self, using the toilet, taking medications, and not bedridden.



- A PCS result is defined as an abnormal laboratory assay result marked as clinically significant in the Investigator's opinion.
- A PCI result is defined as a laboratory assay result that meets criteria tested against as used by the local laboratory for identifying as PCI.

The following subject safety laboratory result items are planned to be listed using the SAS for both protocol parts:

- Chemistry
- Hematology
- Urinalysis
- Drug and Alcohol Screening
- Abnormal results
- PCS results
- PCI results

The following local laboratory result items are planned for table presentation, by treatment groups for each applicable visit using the SAS:

- Chemistry:
  - CFB with descriptive statistics
  - Shift from Baseline with summary statistics
- Hematology:
  - CFB with descriptive statistics
  - Shift from Baseline with summary statistics
- Urinalysis:
  - o CFB with descriptive statistics for numeric results
  - Qualitative summary of Urinalysis
- PCI laboratory results as tested against local laboratory criteria set (see Appendix IV: Potentially Clinically Important Values for list of criteria)
- Marked abnormalities, including the following criteria:
  - $\circ$  Alanine aminotransferase (ALT) > 1.5 x upper limit of normal (ULN)
  - o Bilirubin > 1.5 x ULN (where if fractioned, direct bilirubin >= 35%)
  - ALT or aspartate aminotransferase (AST) > 3 x ULN and total bilirubin (TBL) > 2
     x ULN and alkaline phosphatase (ALP) > 1.5 x ULN (Hy's law)

A list of local laboratory assays planned to be performed can be found in Appendix III:Appendix III:Summary of Laboratory Assays Performed. The planned timings of laboratory sample collection are given in Appendix I: Schedule of Assessments and Procedures.






The following ECG listings will be presented for both protocol parts using the SAS:

- Quantitative results containing all the measurements listed in Table 3.
- Potentially clinically significant results.

The following ECG summary tables are planned, by treatment groups using the SAS:

- CFB with descriptive statistics on all the measurements listed in Table 3.
- Categorical Outliers and marked abnormalities, including the following criteria:

For marked abnormalities:

- o QTcB > 450 (msec) for male subjects.
- $\circ$  QTcB > 470 (msec) for female subjects.
- o Increase in QTcB from baseline  $\geq$  60 (msec).
- o Increase in heart rate CFB%  $\geq$  30% AND observed heart rate  $\geq$  90 (bpm).

For categorical outliers:

- $\circ$  QTcB > 500 (msec).
- o Increase in QTcB from baseline  $\geq 30$  (msec) and < 60 (msec).
- o Increase in QTcB from baseline  $\geq$  60 (msec).
- Time-matched, placebo-adjusted QTcB CFB for all post-dose timepoints ≤ 24 hours.

The following figures are planned for presentation ECG parameter QTcB for both parts of study by treatment groups using the SAS:

- Mean observed values after study drug infusion on dosing days (by dose group)
- Mean observed values over time (excluding post-dose assessments on dosing days)
- Mean CFB after study drug infusion on dosing days (by dose group)




- Mean CFB over time (excluding post-dose assessments on dosing days)
- Placebo-corrected mean CFB in QTcB with 90% CI whiskers across post-dose timepoints up to 24 hours (by dose group)

A time-matched analysis of change in QTcB will be graphically explored. The mean CFB in QTcB versus placebo will be plotted at the different timepoints ≤ 24 hours post-dose, along with 90% 2-sided CI. The upper limit of the 90% CI should be below the 10 (msec) bound as provided by the International Conference on Harmonization (ICH) E14 guideline to be deemed as having no QTc prolongation effect. Due to the small number of subjects planned per cohort, subjects from the different cohorts will be pooled into active treatment and placebo. If any upper limits are observed above the 10 (msec) mark from the pooled plot, further exploration by cohort may be explored. The estimates and 90% CI will be obtained through an analysis of covariance (ANCOVA), using baseline QTcB as covariate and treatment (pooled active and placebo) as effect.

The following example SAS® code can be utilized and modified as needed:

```
Proc GLM Data = <Dataset>;
    By <Tmpt>;
    Class <TRT>;
    Model <CFB> = <TRT> <BaseVal> / solution;
    LSmeans <TRT> / diff cl Alpha = 0.1 pdiff;
    ods output LSMeanDiffCL = <estmt>;
    Run;
Quit;
```

Where <Dataset> is the input dataset, <Tmpt> is the timepoint, <TRT> if is the treatment group, <BaseVal> is the baseline value and <estmt> is the output set containing the estimate and corresponding 90% CI.

The data for these presentations will obtained from the following eCRFs:

- 12-Lead Electrocardiogram Details.
- Vital Signs (for heart rate).

Table 3 below gives the ECG measurements to be assessed.

Table 3. ECG Measurements

| Measurement |
|---------------------------------------------------------------|
| QT interval (msec) |
| QT, corrected with Bazett's formula<br>(QTcB) interval (msec) |
| QRS interval (msec) |
| PR interval (msec) |
| Heart Rate (HR) (bpm) |

The planned timings of these ECG are given in Appendix I: Schedule of Assessments and Procedures.




# 12.4. VITAL SIGNS

Listings will be presented on the following vital sign items separately for both protocol parts using the SAS:

- Quantitative results on all the tests listed in Table 4.
- Potentially clinically significant results (Refer marked abnormalities listed under).

The following vital sign tables are planned to be presented, by treatment groups using the SAS:

- CFB with descriptive statistics on all the tests listed in Table 4.
- Marked abnormalities including the following criteria:
  - Decrease in systolic blood pressure (SBP) of ≥ 25 (mmHg) versus baseline (orthostatic hypotension).
  - Decrease in diastolic blood pressure (DBP) of ≥ 15 (mmHg) versus baseline (orthostatic hypotension).
  - o Increase/decrease in SBP of  $\geq 20$  (mmHg) versus baseline.
  - o Increase/decrease in DBP of  $\geq$  10 (mmHg) versus baseline.
  - o Increase/Decrease in Weight of  $\geq$  7% versus baseline.
  - o Increase/Decrease in Heart Rate by 15 bpm.

The data for these presentations will be obtained from the following eCRFs:

- Vital Signs.
- Physical Examination (for weight).

Table 4 below gives the vital sign tests to be performed.

Table 4. Vital Sign Tests Performed

| Test |
|--------------------------------------|
| Pulse (bpm) |
| Pulse oximetry, SPO <sub>2</sub> (%) |
| Respiratory rate (brpm) |
| Supine DBP (mmHg) |
| Supine SBP (mmHg) |
| Temperature (°C) |
| Weight (kg) |

The planned timings for the vital signs measurements are given in Appendix I: Schedule of Assessments and Procedures.

# 12.5. COLUMBIA SUICIDE SEVERITY RATING SCALE

The Columbia Suicide Severity Rating Scale (C-SSRS) will be listed for both protocol parts separately using the SAS.


The information for these presentations will be obtained from the following eCRFs:

- C-SSRS Screening
- C-SSRS Since Last Visit

The C-SSRS responses over time will be tabulated using count and percent by treatment groups throughout the study, using SAS.

# 13.OTHER RELEVANT DATA ANALYSES/SUMMARIES

# 13.1. HOSPITALIZATIONS AND CLINICAL UNIT CONFINEMENT

A combined listing on the following items will be presented using the SAS separately for both protocol parts:

- Hospitalizations
- Clinical unit confinement

The information for these presentations will be obtained from the following eCRFs:

- Adverse Events Details eCRF
- Clinical Unit Confinement

Duration per hospital stay is calculated in days as:

 $Hospitalization\ Duration\ (days) = (Discharge\ Date-Admission\ Date) + 1$ 

Duration of clinical unit confinement is calculated in days as:

Clinical Unit Confinement Duration (days) = (Discharge Date – Admission Date) + 1

It should be noted that the above duration definitions consider part of a day to count as a whole day.

# 13.2. PHYSICAL AND NEUROLOGICAL EXAMINATIONS

A listing of physical and neurological examination findings for both protocol parts will be presented separately using the SAS.

The information for the listing will be obtained from the following eCRFs:

- Physical and Neurological Examination
- Physical and Neurological Exam Abnormalities

It should be noted that weight will be presented and summarized alongside the vital signs (see Section 12.4 for details), and height will be presented alongside demographics and baseline characteristics (see Section 10.2 for details).

Body systems to assess include:




- Cardiovascular
- Respiratory
- Gastrointestinal
- Neurological (Mental status, Motor and Sensory Skills, Hearing and Speech, Vision, Coordination, Balance)

#### **13.3.IMMUNOGENICITY ANALYSIS**

To assess the immunogenicity of TB006, the presence of anti TB006 antibodies, and associated titer values will be listed by patient and time point for both protocol parts using SAS.

The anti-drug antibody titer values will be summarized descriptively for all subjects, by treatment groups and baseline AD severity stratifications (for Part 2 only), using SAS. Also, the status of anti-drug antibody will be tabulated by treatment groups and baseline AD severity stratifications (for Part 2 only), using SAS.

#### 14.REFERENCES

- 1. ICH E3: Structure and Content of Clinical Study Reports, CDER, FDA (1996).
- 2. ICH E9: Statistical Principles for Clinical Trials, CDER, FDA (1998).
- 3. TB006AD2102 MAD Protocol V3 Am2 Docusign 15Oct2021.
- 4. TB006AD2102 eCRF Specification v2.0 09NOV2021 Final
- 5. TRU212572 CDR System Statistical Analysis Plan V2.0 13 Jan 2022.




### 15.APPENDICES

# Appendix I: SCHEDULE OF ASSESSMENTS AND PROCEDURES

Table 5. Part 1 - Schedule of Activities

| | -2ª | | | | | | St | udy I | Drug | Adm | inistr | ation | Per | iod | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D -28 to D -2 | D -2ª | D-1ª | DIa | D2-6ª | D8 | D9-13a | D15ª | D16-20a | D22a | D23-27 <sup>a</sup> | D29a | D30-34ª | D36ª | D64a | D104ª | E/D <sub>b</sub> | |
| | | | | <b>*</b> | h | li. | Gene | ral a | nd Sa | fety. | Asses | ssmei | nts | de: | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | | |
| Eligibility criteria | X | | X | | | | | | | | | | | | | | | Recheck eligibility before<br>randomization and/or first dose of<br>study drug |
| Medical history <sup>c</sup><br>(includes substance<br>usage) | X | X | х | | | | | | | | | | | | | | | Medical occurrences that begin<br>before the start of study drug but<br>after obtaining informed consent<br>will be recorded on the Medical<br>History/Current Medical Conditions<br>section of the CRF, not the AE<br>section |
| Demography | X | | | | | | | | | | | | | | | | | |
| Physical and<br>neurological<br>examination | X | | х | | | | | | | | | | | X | | X | X | Physical examination will include<br>height (screening only) and weight<br>measurements; see also Section<br>8.2.1 of Protocol |
| Randomization | | | X | 0 | 6 G | | | | | | 8 | | | | | | | |
| Vital signs | x | | X | X | | x | | X | | X | | X | | X | X | X | X | Pre-dose, then 2 and 6 hours after<br>the end of the study drug infusion<br>on D1, D8, D15, D22, D29;<br>otherwise once on the days<br>indicated; see Section 8.2.2 of<br>Protocol for vital signs assessments |




Table 5. Part 1 - Schedule of Activities

| | 2. | | | | | | St | udy I | Drug | Adm | inistr | ation | Per | iod | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2ª | | D -1a | DIa | D2-6ª | D8 | D9-13 <sup>a</sup> | D15a | D16-20a | D22ª | D23-27 <sup>a</sup> | D29a | D30-34 <sup>a</sup> | D36 a | D64ª | D104a | E/D <sub>b</sub> | |
| 12-lead ECG | х | | Х | Х | | X | | X | | X | | X | | X | X | х | X | D1, D8, D15, D22, D29: pre-dose, then 2 and 6 hours after end of study drug infusion D-1, D36, D64, D104, E/D: time-matched with D1, D8, D15, D22, D29 pre-dose to the extent possible |
| AE monitoring | | | | X | х | X | X | X | X | X | X | X | X | X | X | X | X | All AEs and SAEs will be collected from the time of the first study drug administration until D104. |
| Prior/concomitant<br>medication review | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| C-SSRS | X | | | X | | X | | X | | X | | X | | X | X | X | X | |
| Clinical unit confinement | | X | х | х | | X | | X | | X | | X | | | | | | At least 6 hours following study drug administration on dosing days; discharge from the clinical unit will be at the discretion of the investigator provided there are no safety concerns identified from review of the clinical data. Optional overnight confinement from either D -2 or D -1 and on days prior to other dosing days (D7, D14, D21, D28) |
| Outpatient visit | | | X | | | | | | | | j. | | | X | Х | X | X | If the patient is not overnight confined on D -1 (see above), the D -1 visit will be an outpatient visit |




Table 5. Part 1 - Schedule of Activities

| | .2ª | | | | | | St | udy I | Orug | Adm | inisti | ation | Peri | iod | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2a | D -2ª | D -1ª | DIª | D2-6ª | D8 | D9-13a | D15a | D16-20a | D22ª | D23-27 <sup>a</sup> | D29a | D30-34a | D36 a | D64 <sup>a</sup> | D104a | E/D <sub>b</sub> | |
| Site to contact patient | | | | | Х | | X | | X | | X | | X | | | | | Investigator or designee to telephone the patient between D2-6, D9-13, D16-20, D23-27, and D30-34 |
| | | | | | | | Centi | al La | abora | tory | Asse | ssme | nts | | | | | |
| Viral serology (HBsAg,<br>IGM anti-HBe,<br>anti-HCV, HIV) and<br>COVID-19 | X | | | i. | | | | | 100 | | | | | | AG<br>SI | | | |
| Urine alcohol | X | | X | · · | | | | | | | | X | | X | | | | Locally performed at site |
| Drug screening | X | | X | | | | | | | | | X | | X | | | | |
| Clinical laboratory tests<br>(clinical chemistry,<br>hematology, urinalysis) | X | | X | | | X | | | | X | | | 2.3 | X | | X | X | |
| | | | Phari | macod | lynai | nic A | Lssess | men | ts: Co | ogniti | on T | estin | g, MI | RI, BI | lood ! | Samp | les | |
| MMSE | X | | X | | | | | X | | | | | | X | X | X | X | |
| Clinical Dementia<br>Rating scale | | | X | | | | | X | | | | | | X | X | X | X | |
| Cognitive Drug<br>Research Dementia<br>Rating battery <sup>d</sup> | X | | X | | | X | | X | | X | | X | | X | X | X | X | |
| NPI | | | X | | | | | | | | | | | X | X | X | X | |
| Blood sample for PD assessment | | Ī | X | 1 | | | | | | | | | | X | | X | X | Fluid biomarkers will be determined in plasma |
| | | | | | | | | Sti | udy 1 | reati | nent | | | | | | | |
| Study drug IV infusion | | | | X | | X | | X | | X | | X | | | | | | |


TrueBinding
11Apr2022

Table 5. Part 1 - Schedule of Activities

| | -2ª | | | | | | St | udy I | rug | Adm | inistr | ation | Peri | od | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2 | D -2ª | D -1ª | D1ª | D2-6ª | D8 | D9-13a | D15a | D16-20ª | D22ª | D23-27 <sup>a</sup> | D29a | D30-34ª | D36 a | D64ª | D104a | E/D <sub>b</sub> | |
| * | | | | | | - | | Ph | arma | cokir | etics | | | S. | | | | |
| Blood sample for PK assessment | | | | X | | X | | | | | | X | | X | X | X | X | Pre-dose, end of infusion, then 1, 2, 4, and 6 hours after the end of infusion on D1, D8, and D29; single time point on other days |
| Blood sample for ApoE4 genotyping | X | | | | 33 | \$1 | | | | | | | | | | | | Optional ApoE4 sampling is<br>collected at screening but can be<br>taken at any visit until the last study<br>visit (Section 8.7 of Protocol) |
| | | | | | 1 | Phar | maco | kinet | ics aı | nd Ph | arma | acody | nam | ics | | | | |
| Blood sample for ADA assessment | | | | X | | X | | | | | | | | X | | X | | ADA assessment is performed on<br>blood sample collected for PK<br>assessments; D1 and D8 assessment<br>is performed on the pre-dose sample |
| Lumbar puncture for<br>CSF collection <sup>e</sup> | | | Х | | | | | | | | | | | X | | | | Lumbar puncture indicated for D-1<br>can be performed any time between<br>D-8 and D-1<br>CSF biomarkers, and TB006 levels<br>will be determined in CSF |

AD = Alzheimer's Disease; ADA = anti-drug antibody; AE = adverse event; anti-HCV = hepatitis C virus antibody;

ApoE4 = apolipoprotein E4; COVID = coronavirus disease; CRF = case report form; C-SSRS = Columbia Suicide Severity Rating Scale; CSF = cerebrospinal fluid; D = Day; DSM-5 = Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition; ECG = electrocardiogram; E/D = Early Discontinuation; HBsAg = hepatitis B surface antigen; IgM anti-HBc = immunoglobulin M antibody to hepatitis B core antibody; IV = intravenous(ly); MMSE = Mini-Mental State Examination; NINCDS-ADRDA = National Institute of Neurological and Communicative Disorders and Stroke – Alzheimer's Disease and Related Disorders Association; NPI = Neuropsychiatric Inventory; PD = pharmacodynamic(s);

PK = pharmacokinetic(s); SAE = serious adverse event.

Visit days and procedures are allowed a window of  $\pm 2$  days from Day 1 to End of Treatment.

b Applicable only for patients who discontinue early from the study.


Statistical Analysis Plan: TB006AD2102



c The medical history assessed at the screening visit should include prior AD treatment assessment(s). Establishing the clinical diagnosis of AD should include use of criteria from the DSM-5 – Criteria for Major Neurocognitive Disorder (previously dementia) (Section 10.4 of Protocol, Appendix 4) and the NINCDS-ADRDA (Note: ADRDA is now the Alzheimer's Association) (Section 10.5 or Protocol, Appendix 5).

- d The Cognitive Drug Research battery is to be performed twice during the screening visit in both Part 1 and Part 2.
- e The lumbar puncture procedure is optional.




| | .2ª | | | | | | St | udy I | rug | Adm | inistr | ation | Peri | iod | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2a | D -2ª | D -1a | DIa | D2-6ª | D8 | D9-13a | D15a | D16-20a | D22ª | D23-27a | D29a | D30-34ª | D36 a | D64ª | D104ª | E/Db | |
| | | | | | | | Gene | ral an | ıd Sa | fety A | Asses | smen | ts | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | | |
| Eligibility criteria | Х | | X | | | | | | | | | | | | | | | Recheck eligibility before<br>randomization and/or first dose of<br>study drug |
| Medical history <sup>c</sup><br>(includes substance<br>usage) | X | X | X | | | | | | | | | | | | | | | Medical occurrences that begin<br>before the start of study drug but<br>after obtaining informed consent<br>will be recorded on the Medical<br>History/Current Medical<br>Conditions section of the CRF, not<br>the AE section |
| Demography | X | | | | | | | | | | | | | | | | | |
| Physical and<br>neurological<br>examination | X | | X | | | | | | , | | | | | X | | X | X | Physical examination will include<br>height (screening only) and weight<br>measurements; see also Section<br>8.2.1 of Protocol. |
| Randomization | | | X | | | | | | | | | | | | | | | |
| Vital signs | X | | X | X | | X | | x | | x | | X | | х | X | X | X | Pre-dose, then 2 and 6 hours after<br>the end of the study drug infusion<br>on D1, D8, D15, D22, D29;<br>otherwise once on the days<br>indicated; see Section 8.2.2 of<br>Protocol for vital signs assessment |




| | .2ª | | | | | | St | udy I | rug | Adm | inistr | ation | Per | iod | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2ª | D -2ª | D -1a | DIa | D2-6 <sup>a</sup> | D8 | D9-13a | D15a | D16-20a | D22ª | D23-27a | D29a | D30-34a | D36 a | D64ª | D104ª | E/D <sup>b</sup> | |
| 12-lead ECG | X | | X | х | | X | | X | | X | | X | | Х | | X | Х | D1, D8, D15, D22, D29: pre-dose, then after end of study drug infusion D-1, D36, D104, E/D: time-matched with D1, D8, D15, D22, D29 pre-dose to the extent possible |
| AE monitoring | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | All AEs and SAEs will be collected from the time of the first study drug administration until D104. |
| Prior/concomitant<br>medication review | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| C-SSRS | X | | | X | | X | | X | | X | | X | | X | X | X | X | |
| Clinical unit confinement | | х | X | х | | x | | x | | x | | x | | | | | | At least 6 hours following study drug administration on dosing days; discharge from the clinical unit will be at the discretion of the investigator provided there are no safety concerns identified from review of the clinical data. Optional overnight confinement from either D -2 or D -1 and on days prior to other dosing days (D7, D14, D21, D28) |
| Outpatient visit | | | Х | | | | | | | | | | | X | X | X | X | If the patient is not overnight confined on D -1 (see above), the D -1 visit will be an outpatient vis |




| | a a | | | | | | Sti | udy D | )rug | Adm | inistr | ation | Peri | iod | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2a | D -2ª | D -1ª | D1ª | D2-6ª | D8 | D9-13a | D15a | D16-20a | D22ª | D23-27 <sup>a</sup> | D29a | D30-34 <sup>a</sup> | D36 a | D64ª | D104ª | E/Db | |
| Site to contact patient | | | | | X | | x | | X | | X | | X | | | | | Investigator or designee to telephone the patient between D2-6, D9-13, D16-20, D23-27, and D30-34 |
| | | | | | | ( | Centr | al La | bora | tory | Asses | smen | its | | | | | |
| Viral serology (HBsAg,<br>IGM anti-HBe,<br>anti-HCV, HIV) and<br>COVID-19 | X | _ | | | . 0 | 2 | | | | | | | | | | | | |
| Urine alcohol | X | | X | | | | | | | | 5 | X | | X | | | | Locally performed at site |
| Drug screening | X | | X | | | | | | | | | X | | X | | | | |
| Clinical laboratory tests<br>(clinical chemistry,<br>hematology, urinalysis) | X | | X | | | X | | | | X | | | | X | | X | X | |
| | | | Pharr | nacod | ynan | nic A | ssess | ments | s: Co | gnitie | on Te | sting | , MR | I, Bl | ood S | ampl | es | |
| MMSE | X | | X | | | | | X | | | | | | X | X | X | X | |
| Clinical Dementia<br>Rating scale | | | X | | | | | X | | | | | | X | X | X | X | |
| Cognitive Drug<br>Research System<br>battery <sup>d</sup> | X | | X | | | X | | X | | X | | X | | X | X | X | X | |
| NPI | | | X | | | | | | , and | | | | | X | X | X | X | |
| Blood sample for PD assessment | 5 | | X | | | 8 | | | 23<br>5 - 93 | | | 3 - 5 | | X | | X | X | Fluid biomarkers will be<br>determined in plasma |
| | | | | | | | | Stu | dy T | reatn | nent | | | | | | | |
| Study drug IV infusion | | | | X | | X | | X | | X | | X | | | | | | |




| Table 6. Part 2 - Sch | | of Ac | tiviti | es | | | St | ndv I | ) mag | Adm | inicts | etior | Pori | od | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-2ª | D -2ª | D -1ª | DIa | D2-6ª | D8 | D9-13ª | D15a | D16-20ª | D22ª | ex | | D30-34ª | D36 " | D64ª | D104ª | E/Db | Notes |
| | | | | W- | | | | Pha | rma | cokin | etics | | | | - | | | |
| Blood sample for PK assessment | | | | X | | | | | | | | X | | X | X | X | X | Pre-dose and the end of infusion on<br>D1 and D29; single sample on<br>other days |
| Blood sample for ADA assessment | | | | х | | | | | | | | | | X | | x | | ADA assessment is performed on<br>blood sample collected for PK<br>assessments; D1 assessment is<br>performed on the pre-dose sample |
| Blood sample for ApoE4 genotyping | X | | | | | | | | | | | | | | | | | Optional ApoE4 sampling is<br>collected at screening but can be<br>taken at any visit until the last<br>study visit (Section 8.7 of Protocol) |

AD = Alzheimer's Disease; ADA = anti-drug antibody; AE = adverse event; anti-HCV = hepatitis C virus antibody;

ApoE4 = apolipoprotein E4; COVID = coronavirus disease; CRF = case report form; C-SSRS = Columbia Suicide Severity Rating Scale; D = Day; DSM-5 = Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition; ECG = electrocardiogram; E/D = Early Discontinuation; HBsAg = hepatitis B surface antigen; IgM anti-HBc = immunoglobulin M antibody to hepatitis B core antibody; IV = intravenous(ly); MMSE = Mini-Mental State Examination;

NINCDS-ADRDA = National Institute of Neurological and Communicative Disorders and Stroke – Alzheimer's Disease

and Related Disorders Association; NPI = Neuropsychiatric Inventory;

europsychiatric Inventory; PD = pharmacodynamic(s);

PK = pharmacokinetic(s); SAE = serious adverse event.

- a Visit days and procedures are allowed a window of  $\pm 2$  days from Day 1 to End of Treatment.
- b Applicable only for patients who discontinue early from the study.
- c The medical history assessed at the screening visit should include prior AD treatment assessment(s). Establishing the clinical diagnosis of AD should include use of criteria from the DSM-5 Criteria for Major Neurocognitive Disorder (previously dementia) (Section 10.3 of Protocol, Appendix 4) and the NINCDS-ADRDA (Note: ADRDA is now the Alzheimer's Association) (Section 10.4 of Protocol, Appendix 5).
- d The Cognitive Drug Research battery is to be performed twice during the screening visit in both Part 1 and Part 2.


Statistical Analysis Plan: TB006AD2102



Appendix II: SUMMARY OF EFFICACY ANALYSES

| CDRS – Sum of Boxes total EAS2 MMRM Part score CDRS – Proportion of EAS2 CMH Part respondent MMSE score EAS2 MMRM Part | |
|---|---|
| score CDRS – Proportion of EAS2 CMH Part respondent | |
| score CDRS – Proportion of EAS2 CMH Part respondent | |
| score CDRS – Proportion of EAS2 CMH Part respondent | |
| respondent | <del></del> |
| MMSE score EAS2 MMRM Part | Secondary analysis |
| | Secondary analysis |
| NPI score EAS2 MMRM Part | Secondary analysis |
| CDRS EAS2 Descriptive statistics Part | Secondary analysis |
| CDRS – Proportion of EAS2 Descriptive statistics Part respondent | Secondary analysis |
| MMSE score EAS2 Descriptive statistics Part | Secondary analysis |
| NPI score EAS2 Descriptive statistics Part | Secondary analysis |




Appendix III: SUMMARY OF LABORATORY ASSAYS PERFORMED

| Laboratory Category | Assay Grouping | Assay |
|---|---|---|
| Chemistry | Electrolytes | Glucose |
| | | Potassium |
| | | Sodium |
| | | Calcium |
| | Renal Function | Blood Urea Nitrogen (BUN) |
| | | Creatinine |
| | Liver Function | Alanine Aminotransferase (ALT) |
| | | Aspartate Aminotransferase (AST) |
| | | Albumin |
| | | Creatine Phosphokinase (CPK) |
| | | Alkaline phosphatase |
| | | Total Bilirubin |
| | | Direct Bilirubin |
| | | Total Protein |
| | Lipid Profile | Total Cholesterol |
| | 2 0 | High-density Lipoprotein (HDL) Cholestero |
| | | Low-density Lipoprotein (LDL) Cholestero |
| | | Triglycerides |
| | | Thyroid-stimulating Hormone (TSH) |
| | | Hemoglobin A1c (HbA1c) |
| Hematology | RBC indices | Platelet count |
| <b></b> | | Red Blood Cell (RBC) count / Erythrocytes |
| | | Hemoglobin |
| | | Hematocrit |
| | | Ery. Mean Corpuscular volume (MCV) |
| | | Ery. Mean Corpuscular Hemoglobin (MCH) |
| | | Leukocytes |
| | White Blood Cell (WBC) Count | Neutrophils Absolute |
| | with differential | Neutrophils Percent |
| | | Lymphocytes Absolute |
| | | Lymphocytes Percent |
| | | Monocytes Absolute |
| | | Monocytes Percent |
| | | Eosinophils Absolute |
| | | Eosinophils Percent |
| | | Reticulocytes Absolute |
| | | Reticulocytes Percent |
| | | Basophils Absolute |
| | | Basophils Percent |
| Urinalysis (dipstick) | 2 | Specific Gravity |
| Ormanysis (aipstick) | | pH |
| | | Glucose |
| | - | Protein |




| Laboratory Category | Assay Grouping | Assay |
|---|---|---|
| | | Occult Blood |
| | | Ketones |
| | | Bilirubin |
| | | Urobilinogen |
| | | Nitrite |
| | | Leukocyte esterase |
| | | Microscopic examination if blood or protein is abnormal |
| Other Screening Tests | Viral serology | Hepatitis B surface antigen (HBsAg) |
| | | IgM Hepatitis B core antibody (anti-HBc) |
| | | Hepatitis C antibody (Anti-HCV) |
| | | Human immunodeficiency virus (HIV) |
| | | COVID19 |
| | Non-childbearing potential only | Follicle-stimulating Hormone (FSH) |
| | | Estradiol |
| | Plasma Alcohol and Urine Blood<br>Screen | Alcohol |
| | 5 | Optiates |
| | | Methadone |
| | 57 | Buprenorphine |
| | | Methamphetamine |
| | 2 | Cocaine |
| | | Amphetamines |
| | WOCBP | Highly sensitive human chorionic-gonatropin (hCG) pregnancy test |




#### Appendix IV: POTENTIALLY CLINICALLY IMPORTANT VALUES

The following table contains a list of ranges used by the laboratory to flag critical laboratory values which will also be used in this study to identify any potentially clinically important values within the table and listings presentations. If a planned laboratory assay does not have applicable PCI criteria limits, that assay is not included in the below table.

| | | | PCI Criteria | Value Limits |
|---|---|---|---|---|
| Laboratory Category | Assay | Unit | Lower | Upper |
| Chemistry | Albumin | g/dL | 2.0 | 6.0 |
| | Alkaline Phosphatase | IU/L | NA | 200 |
| | Alanine Aminotransferase | IU/L | NA | 150 |
| | Aspartate Aminotransferase | IU/L | NA | 150 |
| | Bilirubin | mg/dL | NA | 2.50 |
| | Blood Urea Nitrogen | mg/dL | NA | 30.0 |
| | Calcium | mg/dL | 7.0 | 13.5 |
| | Glucose | mg/dL | 40 | 250 |
| | Potassium | mmol/L | 3.2 | 6.0 |
| | Sodium | mmol/L | 130 | 150 |
| Hematology | Hematocrit (Female) | % | 24.0 | 54.0 |
| | Hematocrit (Male) | % | 24.0 | 60.0 |
| | Hemoglobin (Female) | g/dL | 8.0 | 18.0 |
| | Hemoglobin (Male) | g/dL | 8.0 | 20.0 |
| | Lymphocytes | 0^3/uL | 0.50 | NA |
| | Neutrophils | 0^3/uL | 1.00 | NA |
| | Platelets | 0^3/uL | 75 | 750 |
| | Leukocytes | 0^3/uL | 2.5 | 25.0 |
| Other Screening Tests | Human immunodeficiency virus (HIV) | | Pos | itive |
| | COVID19 | | Pos | itive |
| | Optiates | | Pos | itive |
| | Methadone | | Pos | itive |
| | Buprenorphine | | Pos | itive |
| | Methamphetamine | | Pos | itive |
| | Cocaine | | Pos | itive |
| | Amphetamines | | Pos | itive |


#### **Certificate Of Completion**

Envelope Id: 503598ABA6D14CA8B5F54D0BDEF7031E

Subject: Please DocuSign: TB006AD2102\_SAP\_Ver 2.0\_11Apr2022.docx

Source Envelope:

Document Pages: 50 Certificate Pages: 5

Signatures: 3 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed





#### **Record Tracking**

Status: Original

4/12/2022 3:31:21 AM

Holder:

Location: DocuSign

#### Signer Events

Signature

#### **Timestamp**

Sent: 4/12/2022 3:32:45 AM Viewed: 4/12/2022 3:33:05 AM Signed: 4/12/2022 3:33:41 AM

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signed by link sent to

Signature ID:

053E504E-ECB2-49B9-B7E7-31AE1A775A71

Using

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I am the author of this document

# **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Sent: 4/12/2022 3:32:46 AM Viewed: 4/12/2022 1:06:06 PM Signed: 4/12/2022 1:07:38 PM

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signed by link sent to

Signature ID:

A3EA3B5A-E669-4A04-A339-3E173E8742DB

Using

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure:

Accepted: 4/12/2022 1:06:06 PM

ID: 432114b8-4eda-4a13-ad21-b3fe332c770b

Signer Events

MMS

Security Level: Email, Account Authentication (Required)

**Signature** 

Sent: 4/12/2022 3:32:45 AM Viewed: 4/12/2022 3:47:29 AM Signed: 4/12/2022 3:50:04 AM

**Timestamp** 

Signature Adoption: Pre-selected Style

Signed by link sent to

Signature ID:

CAD557FF-FDB2-4E87-ADA8-0676AEB4ABC2

Using

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I have reviewed this document

Electronic Record and Signature Disclosure: Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered | Hashed/Encrypted Security Checked | 4/12/2022 3:32:46 AM<br>4/12/2022 3:47:29 AM<br>4/12/2022 3:50:04 AM |
| Signing Complete<br>Completed | Security Checked<br>Security Checked | 4/12/2022 1:07:38 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, MMS Holdings Inc. (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact MMS Holdings Inc.:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

#### To advise MMS Holdings Inc. of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at an and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

#### To request paper copies from MMS Holdings Inc.

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with MMS Holdings Inc.

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| required hardware and software | |
|---|---|
| Operating Systems: | Windows2000? or WindowsXP? |
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy<br>Server must enable HTTP 1.1 settings via<br>proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify MMS Holdings Inc. as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by MMS Holdings Inc. during the course of my relationship with you.

Statistical Analysis Plan: TB006AD2102



# ADDENDUM TO STATISTICAL ANALYSIS PLAN: TB006AD2102 FINAL VERSION 2.0 DATED 11 APRIL 2022

**Study Title:** A Seamless Phase 1b/2a Double-blind, Randomized,

Multiple dose, Multi-center, Sequential Doseescalation Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of

TB006 in Patients with Mild to Severe

Alzheimer's Disease

Study Number: TB006AD2102

**Study Phase:** Phase 1b/2a

**Sponsor:** TrueBinding, Inc.

300 Lincoln Center Drive

Suite 200

Foster City, CA, 94404

**Addendum Version:** Final ver 1.0

NCT Number: NCT05074498

**Date:** 14Nov2022

#### **Confidentiality Statement**

This document contains confidential and proprietary information, and is not to be distributed to any third party.




# Table of Contents

| Ad | dendum to Statistical Analysis Plan: TB006AD2102 Final Version 2.0 dated 11 april 2022 | . 1 |
|---|---|---|
| 1. | Signature Page | . 3 |
| 2. | Purpose | . 4 |
| | Descriptions of Changes in Study Conduct and Analysis Planned in Protocol and Statistical Analysis Plan | |
| 4. | References | . 6 |




### 1. SIGNATURE PAGE

**Study Title:** A Seamless Phase 1b/2a Double-blind, Randomized,

Multiple dose, Multi-center, Sequential Dose-escalation

Study to Assess the Safety, Tolerability,

Pharmacokinetics, Pharmacodynamics and Efficacy of

TB006 in Patients with Mild to Severe

Study Number: TB006AD2102

| | Electronically signed<br>by:<br>Reason: I am the<br>author of this document<br>Date: Nov 14, 2022<br>13:41 GMT+5.5 | |
|---|---|---|
| Prepared by: | | Date: |
| | , PhD<br>Principal Biostatistician, Biometrics<br>MMS Holdings, Inc | |
| Reviewed by | Electronically signed by: Reason: I approve this document Date: Nov 14, 2022 18:23 GMT+2 Senior Biostatistician II, Biometrics MMS Holdings, Inc | Date: |
| Approved by | Electronically signed<br>by:<br>PharmD<br>Reason: I approve<br>this document<br>Date: Nov 14, 2022 | Date: |




#### 2. PURPOSE

The Statistical Analysis Plan (SAP) version 2.0 dated 11 April 2022 need to clarify the definition of Efficacy Analysis Set-Part 2 (EAS2). The EAS2 is defined in SAP as:

The Part 2 – Efficacy Analysis Set (EAS2) includes all subjects who received assigned dose of TB006 in Part 2 and the subjects enrolled at the same TB006 dose level in Part 1, as well as all placebo patients will be included and have at least one post-dose evaluable PD assessment across subject.

Here "PD assessment" can be mistaken to refer to plasma or imaging biomarkers and hence the definition for EAS2 is clarified in addendum SAP to replace text "PD" with text "efficacy". The updated definition is as under:

The Part 2 – Efficacy Analysis Set (EAS2) includes all subjects who received assigned dose of TB006 in Part 2 and the subjects enrolled at the same TB006 dose level in Part 1, as well as all placebo patients will be included and have at least one post-dose evaluable **efficacy** assessment across subject.




# 3. DESCRIPTIONS OF CHANGES IN STUDY CONDUCT AND ANALYSIS PLANNED IN PROTOCOL AND STATISTICAL ANALYSIS PLAN

This change will <u>only</u> impact the analysis population definition in SAP version 2.0 dated 11 April 2022, Section 7.1.5.


Statistical Analysis Plan: TB006AD2102



## 4. REFERENCES

1. TrueBinding TB006AD2102 Statistical Analysis Plan Version 2.0 Final signed, dated 11 April 2022.

